CLINICAL TRIAL: NCT02455674
Title: Weight Estimation of A Child With Unknown Age and Height: Using Mean Ages on Clothing Size Labels in Revised APLS Formulas for Weight Estimation. A Prospective Cross-Sectional Study
Brief Title: Using Mean Ages on Clothing Size Labels in Revised Advanced Pediatric Life Support Formulas for Weight Estimation
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: AntalyaTRH003
Record Dates: First submitted 2015-05-21; First posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Body Weight
Keywords: weight estimation; emergency; child
MeSH Terms: conditions — Body Weight; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Age under 6 years: All children 1 to 6 years
  Used formula for weight calculation:
  Children 1-5 years: Weight (kg) = (2 × age in years) + 8
- Age over 6 years: All children 6 to 12 years
  Used formula for weight calculation:
  Children 6-12 years: Weight (kg) = (3 × age in years) + 7

SUMMARY:
Weight calculation based on age could be performed according to APLS (Advanced Pediatric Life Support) guideline recommendations in children requiring emergency treatment and intervention in the field or during resuscitation with no active weight and height measurements. The aim of the study is to investigate the suitability of weight calculation using mean ages on clothing size labels (ACL) to the actual weight in real emergencies with no known actual age of the patient (AA).

DETAILED DESCRIPTION:
Weight calculation based on age could be performed according to APLS guideline recommendations in children requiring emergency treatment and intervention in the field or during resuscitation with no active weight and height measurements. Age formulas require only knowledge of the actual age of the child and widely used all over the world with being catchy. However, situations in which one has to intervene a child without having any patient data, including information on children's ages, especially in the field or during resuscitation are not uncommon. The objective of this study is to investigate the availability of age information contained in clothing size labels of children in weight calculation according to APLS recommendations. Usability of labels can protect victims from overdose and underdose problems in cases where the actual age is unknown and the measurements cannot be done

ELIGIBILITY:
Inclusion Criteria:

* All patients between 1-12 years of age who presented to the emergency department and agreed to participate in the study were consecutively included in the study

Exclusion Criteria:

* Age under 1 years and over 12.99 years
* No weighing in ED
* No clothing size label information
* Refused to participate

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Data of children, aged between 1 to 12 years, were consecutively collected. Patients were divided into two groups as under the age of 6 (age <6) and over 6 years of age (age≥6).
Sampling Method: Non-Probability Sample
Enrollment: 1094 (Actual)
Dates: Start 2014-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Correlation of children's actual age and age information on clothing size labels. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Can K Akyol, MD, Study Director — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Department of Emergency, Antalya, Turkey (Türkiye)

REFERENCES:
- [Background] Young TP, Washington O, Flanery A, Guptill M, Reibling ET, Brown L, Barcega B. Comparison of the finger counting method, the Broselow tape and common weight estimation formulae in Filipino children after Typhoon Haiyan. Emerg Med Australas. 2015 Jun;27(3):239-44. doi: 10.1111/1742-6723.12382. Epub 2015 Mar 26. PMID 25818595
- [Background] Graves L, Chayen G, Peat J, O'Leary F. A comparison of actual to estimated weights in Australian children attending a tertiary children's' hospital, using the original and updated APLS, Luscombe and Owens, Best Guess formulae and the Broselow tape. Resuscitation. 2014 Mar;85(3):392-6. doi: 10.1016/j.resuscitation.2013.11.024. Epub 2013 Dec 7. PMID 24321321
- [Background] Sanghera N, Chan PY, Khaki ZF, Planner C, Lee KK, Cranswick NE, Wong IC. Interventions of hospital pharmacists in improving drug therapy in children: a systematic literature review. Drug Saf. 2006;29(11):1031-47. doi: 10.2165/00002018-200629110-00003. PMID 17061909
- [Background] Wells M, Coovadia A, Kramer E, Goldstein L. The PAWPER tape: A new concept tape-based device that increases the accuracy of weight estimation in children through the inclusion of a modifier based on body habitus. Resuscitation. 2013 Feb;84(2):227-32. doi: 10.1016/j.resuscitation.2012.05.028. Epub 2012 Jul 13. PMID 22796544
- [Background] Argall JA, Wright N, Mackway-Jones K, Jackson R. A comparison of two commonly used methods of weight estimation. Arch Dis Child. 2003 Sep;88(9):789-90. doi: 10.1136/adc.88.9.789. No abstract available. PMID 12937099
- [Background] Kelly AM, Nguyen K, Krieser D. Validation of the Luscombe weight formula for estimating children's weight. Emerg Med Australas. 2011 Feb;23(1):59-62. doi: 10.1111/j.1742-6723.2010.01351.x. Epub 2010 Dec 6. PMID 21134132
- [Background] Luscombe MD, Owens BD, Burke D. Weight estimation in paediatrics: a comparison of the APLS formula and the formula 'Weight=3(age)+7'. Emerg Med J. 2011 Jul;28(7):590-3. doi: 10.1136/emj.2009.087288. Epub 2010 Jul 20. PMID 20659877
- [Background] Thompson MT, Reading MJ, Acworth JP. Best Guess method for age-based weight estimation in paediatric emergencies: validation and comparison with current methods. Emerg Med Australas. 2007 Dec;19(6):535-42. doi: 10.1111/j.1742-6723.2007.01031.x. PMID 18021106
- [Background] van Furth R, Braat AG, Leijh PC, Klein F. Opsonic activity and composition of five intramuscular gammaglobulin preparations. J Infect. 1986 Nov;13(3):269-75. doi: 10.1016/s0163-4453(86)91256-9. PMID 2432132
- [Background] Sinha M, Lezine MW, Frechette A, Foster KN. Weighing the pediatric patient during trauma resuscitation and its concordance with estimated weight using Broselow Luten Emergency Tape. Pediatr Emerg Care. 2012 Jun;28(6):544-7. doi: 10.1097/PEC.0b013e318258ac2e. PMID 22653453
- [Background] Lim CA, Kaufman BJ, O'Connor J Jr, Cunningham SJ. Accuracy of weight estimates in pediatric patients by prehospital Emergency Medical Services personnel. Am J Emerg Med. 2013 Jul;31(7):1108-12. doi: 10.1016/j.ajem.2013.04.018. Epub 2013 May 21. PMID 23706580
- [Background] Elgie LD, Williams AR. Using age on clothes size label to estimate weight in emergency paediatric patients. Eur J Emerg Med. 2012 Oct;19(5):338-40. doi: 10.1097/MEJ.0b013e328355abc2. PMID 22914117
- [Background] Krieser D, Nguyen K, Kerr D, Jolley D, Clooney M, Kelly AM. Parental weight estimation of their child's weight is more accurate than other weight estimation methods for determining children's weight in an emergency department? Emerg Med J. 2007 Nov;24(11):756-9. doi: 10.1136/emj.2007.047993. PMID 17954827
- [Background] Leffler S, Hayes M. Analysis of parental estimates of children's weights in the ED. Ann Emerg Med. 1997 Aug;30(2):167-70. doi: 10.1016/s0196-0644(97)70137-9. PMID 9250640
- [Background] Rosenberg M, Greenberger S, Rawal A, Latimer-Pierson J, Thundiyil J. Comparison of Broselow tape measurements versus physician estimations of pediatric weights. Am J Emerg Med. 2011 Jun;29(5):482-8. doi: 10.1016/j.ajem.2009.12.002. Epub 2010 Apr 2. PMID 20825816
- [Background] Nieman CT, Manacci CF, Super DM, Mancuso C, Fallon WF Jr. Use of the Broselow tape may result in the underresuscitation of children. Acad Emerg Med. 2006 Oct;13(10):1011-9. doi: 10.1197/j.aem.2006.06.042. PMID 17015417
- [Background] Harris M, Patterson J, Morse J. Doctors, nurses, and parents are equally poor at estimating pediatric weights. Pediatr Emerg Care. 1999 Feb;15(1):17-8. doi: 10.1097/00006565-199902000-00005. PMID 10069305
- [Background] Greig A, Ryan J, Glucksman E. How good are doctors at estimating children's weight? J Accid Emerg Med. 1997 Mar;14(2):101-3. doi: 10.1136/emj.14.2.101. PMID 9132182
- [Background] Meguerdichian MJ, Clapper TC. The Broselow tape as an effective medication dosing instrument: a review of the literature. J Pediatr Nurs. 2012 Aug;27(4):416-20. doi: 10.1016/j.pedn.2012.04.009. Epub 2012 May 8. No abstract available. PMID 22579781